CLINICAL TRIAL: NCT05108233
Title: Evaluation of Sleep Quality in Head and Neck Cancer Patients Throughout Treatment Course
Status: Withdrawn | Type: Observational
Why Stopped: PI agreed to close study as prompted by PRMC inquiry
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 21D.668; JT 16663 (Other: JeffTrial Number)
Record Dates: First submitted 2021-10-04; First posted 2021-11-04 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Malignant Head and Neck Neoplasm
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey): COHORT 1-TP1: Patients complete surveys over 20 minutes on post-op day 3 and on day of discharge (or within 1 week).
  COHORT 1-TP2: Patients complete surveys over 15 minutes at all regularly scheduled follow-up appointments (approximately 1 month, 3 months, 6 months, 12 months).
  COHORT 2: Patients complete surveys over 15 minutes once.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Complete survey

SUMMARY:
This study examines how head and neck cancer treatment affects quality of sleep over time and factors that contribute to sleep quality. Sleep plays a critical role in healing and quality of life, and recent studies investigating sleep disorders in head and neck cancer patients reveal sleep quality is a major determinant of post-treatment outcomes. Information from this study may help researchers better understand how treatment impacts sleep quality so that they can make changes that may help improve patient sleep quality.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To describe the five (5) components of sleep quality in head and neck patients under different stages of post-op treatment and different environment.

II. To evaluate the effect of surgery, treatment and environment on the five (5) components of sleep quality in head and neck cancer patients.

SECONDARY OBJECTIVES:

I. To evaluate the association between the five (5) components of sleep quality and comorbid obstructive sleep apnea (STOP-BANG and Epworth Sleeping Scale) and depression (Patient Health Questionnaire-2 [PHQ-2]), under different stages of post-op treatment and different environment.

II. To evaluate the association between Fitbit actigraphy data (i.e. the 5th component of sleep quality) and the first 4 components of sleep quality for inpatients.

III. To compare the inpatient versus the outpatient responses on sleep hygiene at different time points of measurement.

EXPLORATORY OBJECTIVE:

I. To assess whether survey results warrant additional counseling or patient education.

OUTLINE:

COHORT 1-TP1: Patients complete surveys over 20 minutes on post-op day 3 and on day of discharge (or within 1 week).

COHORT 1-TP2: Patients complete surveys over 15 minutes at all regularly scheduled follow-up appointments (approximately 1 month, 3 months, 6 months, 12 months).

COHORT 2: Patients complete surveys over 15 minutes once.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Adult at least 18 years old
* Capable of giving informed consent
* Diagnosed with head and neck cancer (previously untreated, any stage)
* Treatment plan involves surgery
* Willing to comply with all study procedures and be available for the duration of the study
* English-speaking

Exclusion Criteria:

* Non-English speaking
* Pre-existing sleep disorder defined below:

  * Obstructive sleep apnea
  * Insomnia
  * Narcolepsy
  * Restless leg syndrome
  * Rapid eye movement (REM) sleep behavior disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with head and neck cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Time in bed | Up to study completion; approximately 12 months
  The time difference between time to get into bed and time to get up, measured in minutes
Sleep latency | Up to study completion; approximately 12 months
  How long it takes to sleep, measured in minutes.
Number of nighttime awakening | Up to study completion; approximately 12 months
Sleep maintenance latency | Up to study completion; approximately 12 months
  How long it takes to fall back to sleep, measured in minutes.
Per-patient average score on Richards-Campbell Sleep Questionnaire | Up to study completion; approximately 12 months
Sleep hygiene | Up to study completion; approximately 12 months
Barriers to sleep quality | Up to study completion; approximately 12 months
Per-patient sum of scores on Epworth Sleepiness Scale | Up to study completion; approximately 12 months
Per-patient sum of positive responses on STOP-BANG | Up to study completion; approximately 12 months
Per-patient sum of scores on Patient Health Questionnaire-2 | Up to study completion; approximately 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States